CLINICAL TRIAL: NCT05303610
Title: Effects of Tissue Properties of the Superficial Anterior Myofascial Chain on the Development of Patellofemoral Pain Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, research assistant, Istanbul Medeniyet University
Other Study IDs: 2022/0077
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-03

CONDITIONS: Patellofemoral Syndrome; Knee; Connective Tissue; Fascia
Keywords: Patellofemoral Syndrome; knee; connective tissue; fascia
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: This group will consist of 28 patients with diagnosed Patellofemoral pain syndrome, aged between 25-50 years.
  Interventions: Other: Observational
- Control group: Healthy individuals between the ages of 25-50 and without any orthopedic (Anterior cruciate ligament rupture, Meniscal tears etc.), neurological (Multipl sclerosis, Stroke etc) and rheumatological disorders (Rheumatoid arthritis, Ankylosing spondylitis etc.).
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is a cross sectional study. The aim of the study is to evaluate the myofascial chain lines in addition to the general evaluation parameters in patients with patellofemoral pain syndrome (PFPS) and to determine whether deviations from normal in the myofascial structure have an effect on the development of PFPS.

SUMMARY:
The aim of the study is to evaluate the myofascial chain lines in addition to the general evaluation parameters in patients with patellofemoral pain syndrome (PFPS) and to determine whether deviations from normal in the myofascial structure have an effect on the development of PFPS.

There will be two groups in this study. One of the groups will consist of 28 patients aged between 25-50 years. The other group will consist of 28 healthy individuals between the ages of 25-50 years. Postural problems that can be seen in the superficial anterior myofascial chain line will be evaluated. These problems: forward head, q-angle, genu varum, genu valgum, foot postural problems (pes planus, pes kavus vb.) and pelvic tilt. In addition to all these assessments, knee pain and the biomechanical properties of the anterior myofascial tissue will be evaluated.

DETAILED DESCRIPTION:
Although many factors such as lower extremity malalignment, quadriceps muscle weakness, hamstring, gastrocnemius, tensor fascia latae muscle shortness, iliotibial band tension, lower extremity malalignment have been shown to be effective in the development of PFPS, it has been reported in recent studies that these factors which cause patellofemoral pain syndrome may also be related to fascia. The aim of the study is to evaluate the myofascial chain lines in addition to the general evaluation parameters in patients with patellofemoral pain syndrome (PFPS) and to determine whether deviations from normal in the myofascial structure have an effect on the development of PFPS. It was stated that the fascial chain containing the PFPS-related regions is the Superficial Anterior Chain, and this chain starts from the toe extensors and ends at the masteoid process.

There will be two groups in this study. One group of this study will include 28 individuals aged 25-50, diagnosed with PFPS, with pain in the retropatellar region for at least 6 months and non-traumatic. The other group of this study will include 28 healthy individuals between the ages of 25-50 and without any orthopedic (Anterior cruciate ligament rupture, Meniscal tears etc.), neurological (Multipl sclerosis, Stroke etc) and rheumatological disorders (Rheumatoid arthritis, Ankylosing spondylitis etc.).

Postural problems that can be seen in the superficial anterior myofascial chain line will be evaluated. These problems: forward head, q-angle, genu varum, genu valgum, foot postural problems (pes planus, pes kavus vb.) and pelvic tilt. In addition to all these assessments, knee pain and the biomechanical properties of the anterior myofascial tissue will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Patellofemoral pain syndrome,
* Volunteers between the ages of 25-50,
* Having pain in the retropatellar region for at least 6 months that is not a result of trauma,
* Not having received medical treatment and/or physiotherapy for PFPS in the last 6 months.

Exclusion Criteria:

* Having history of lower extremity, pelvis and spine surgery/fracture in the last 6 months,
* Having orthopedic (Anterior cruciate ligament rupture, Meniscal tears, etc), neurological (Multiple sclerosis, paralysis-paralysis, etc.) and/or rheumatological (rheumatoid arthritis, ankylosing spondolitis, etc.) problems,
* Pregnancy ,
* Having a history of connective tissue disease,
* Using sedatives and/or muscle relaxants that may alter muscle tone.

Ages: 25 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Persons who meet the inclusion criteria and who volunteered to participate in the study, who applied to the Orthopaedic outpatient clinic of the Medical Faculty Hospital will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-05-05 (Estimated); Study Completion 2023-06-03 (Estimated)

PRIMARY OUTCOMES:
Knee pain | baseline
  Visual Analogue Scale (VAS) will be used in the assessment of pain severity. VAS expresses pain severity between a score of 0 (no pain) and 10 (unbearably severe pain). The subject is asked to mark the score that best reflects the severity of knee pain he/she feels.
Forward head | baseline
  The end point of the superficial anterior myofascial chain considered in the study is the mastoid process. And to this point attach muscles such as the sternocleidomastoid (SCM) that affect head and neck movements and position. In case of shortness of these muscles, forward tilt of the head may occur. The craniovertebral angle will be considered in determining the forward tilt of the head. In this study, markers will be placed on the mastoid process and C7 spinous process to determine the craniovertebral angle. Photographs of the individual will be taken from the front and side, and then the craniovertebral angle will be calculated using the Tracker 4.11.0 software on these photos. FHP is characterized as pathologic when the craniovertebral angle (CVA) is ≥50°.
Q-Angle | baseline
  For the Q angle, the angle between a straight line from the SIAS to the center of the patella and the line from the center of the patella to the center of the tuberositas tibia will be measured with a goniometer. While the Q angle can be between 6° and 27°, its approximate average value is 15°. Increasing or decreasing the Q angle increases the pressure in the lateral and medial compartments of the patellofemoral joint.
  4- Genu varum
Genu varum | baseline
  The individual in the standing position is asked to unite the lower extremities while maintaining 0° extension of the knees. The distance between the medial condyles is measured as the medial malleolar are in contact. If the distance is more than 1 cm, it indicates the genu varum.
genu valgum | baseline
  The individual in the standing position is asked to unite the lower extremities while maintaining 0° extension of the knees. The distance between the medial malleolar is measured as the medial condyles are in contact. If the distance is more than 1 cm, it indicates the genu valgum.
pes planus | baseline
  Pes Planus will be evaluated with navicular drop test. The distance between the navicular bone and the ground is measured while the individual sits on the chair with the hip-knee joint in 90º flexion and the subtalar joint in neutral position. Then, the distance between the navicular bone and the ground is measured again while the individual is standing in a position with equal weight on both extremities. The difference between the two measurements is recorded. 10 mm or more difference is considered pes planus.
foot posture | baseline
  Foot posture will be evaluated using the Foot posture index, a six item foot posture assessment tool, where each item is scored between -2 and +2 to give a sum total between -12 (highly supinated) and +12 (highly pronated). Items include: talar head palpation, curves above and below the lateral malleoli, calcaneal angle, talonavicular bulge, medial longitudinal arch, and forefoot to rearfoot alignment.
pelvic tilt | baseline
  The position of the pelvis will be evaluated with a digital pelvic inclinometer device to determine whether the pelvis has tilted anteriorly or posteriorly. The digital pelvic inclinometer is a valid and reliable method for the evaluation of pelvic tilt. The device consists of two calipers and the calipers are placed on the SIAS (spina illaca anterior posterior) and SIPS (spina illaca posterior superior) of the pelvis. The score on the digital display is recorded. "-" values indicate posterior pelvic tilt, "+" values indicate anterior pelvic tilt.
Biomechanical and viscoelastic properties of myofascial tissues | baseline
  Biomechanical and viscoelastic properties of myofascial tissues will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). The passive tone and stiffness properties will be calculated by the device from the average of the oscillatory responses of the tissue to this mechanical stimulus. Measurements were taken 3 times from each point and the average values will be used in statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No